CLINICAL TRIAL: NCT05270213
Title: A First-In-Human, Phase 1 a/b Dose Escalation and Expansion Study to Evaluate RBS2418 as Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced Unresectable, Recurrent or Metastatic Tumors
Brief Title: Evaluation of RBS2418 in Subjects With Advanced, Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Riboscience, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBS2418-1001
Record Dates: First submitted 2022-02-09; First posted 2022-03-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer
Keywords: Metastatic tumors; Recurrent tumors; Unresectable tumors
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: The dose escalation phase (Part A) employed a standard 3+3 design to identify dose-limiting toxicities (DLTs), establish the maximum tolerated dose (MTD, if observed), determine dose levels that can achieve Ctrough levels in excess of target inhibition EC90, and determine the recommended doses of RBS2418, both as monotherapy and in combination with pembrolizumab, for further evaluation. The Part A goals have been achieved, and Part A has been completed.
  Part B is in progress to explore the safety and preliminary efficacy of RBS2418 at selected dose levels as monotherapy and in combination with pembrolizumab or other approved anti-cancer therapies.
  Treatment Group A-1: RBS2418 Dose Escalation (Monotherapy) COMPLETED
  Treatment Group A-2: RBS2418 plus Pembrolizumab Dose Escalation (Combination Therapy) COMPLETED
  Treatment Group B: RBS2418 as Monotherapy or in combination with investigator-selected approved anticancer therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A-1 (Completed) (Experimental): For Treatment Group A-1, a cohort of three (3) subjects will be dosed at the starting dose of 100 mg twice a day (BID) of RBS2418. Subsequent subjects will then be enrolled in serial, three (3) subject cohorts, with 100% dose increments (doubling the dose) until 800 mg BID
  Interventions: Drug: RBS2418
- Treatment Group A-2 (Completed) (Experimental): For Treatment Group A-2, a cohort of three (3) subjects will be dosed at the starting dose of 100 mg twice a day (BID) of RBS2418 in combination with pembrolizumab 200 mg IV (administered on Day 1 and every 3 weeks). Subsequent subjects will then be enrolled in serial, three (3) subject cohorts, with 100% dose increments (doubling the dose) until 800 mg BID
  Interventions: Drug: RBS2418; Drug: Pembrolizumab
- Treatment Group B (Experimental): RBS2418 as Monotherapy or in combination with investigator-selected approved anticancer therapy at selected dose levels. (n~140)
  Interventions: Drug: RBS2418; Drug: Pembrolizumab; Drug: Other approved anti-cancer therapy

INTERVENTIONS:
Drug: RBS2418 — RBS2418 is a potent and selective small molecule inhibitor of ectonucleotide pyrophosphatase/phosphodiesterase I (ENPP1). RBS2418 as monotherapy potentially can have an activating effect on the anti-tumor innate immune response and lead to anti-tumor responses in adult subjects with advanced or metastatic tumors.
Drug: Pembrolizumab — 200 mg intravenously every 3 weeks
  Arms: Treatment Group A-2 (Completed); Treatment Group B
Drug: Other approved anti-cancer therapy — Standard of care (SOC) therapy
  Arms: Treatment Group B

SUMMARY:
RBS2418 (investigational product) is a specific immune modulator, working through ectonucleotide pyrophosphatase/phosphodiesterase I (ENPP1), designed to lead to anti-tumor immunity by increasing endogenous 2'-3'-cyclic guanosine monophosphate-adenosine monophosphate (cGAMP) and adenosine triphosphate (ATP levels) and reducing adenosine production in the tumors. RBS2418 has the potential to be an important therapeutic option for subjects both as monotherapy and in combination with other cancer treatments including monotherapy and in combination with other cancer treatments including immunotherapy or chemotherapy. This study is an open-label, multi-site Phase 1a/1b study of RBS2418, a selective ENPP1 inhibitor, in combination with pembrolizumab or other approved anticancer therapies or as a monotherapy in subjects with advanced unresectable, recurrent or metastatic tumors. The phase 1a (dose escalation phase) has been completed. The Phase 1b expansion phase of the study has been increased in size and scope.

DETAILED DESCRIPTION:
The dose escalation phase (Part A) of this Phase 1a/1b study has been completed (n=24 study participants). Based on safety and preliminary activity data, we have expanded the size and scope of the dose expansion phase (Part B), which will include treatment groups receiving RBS2418 at selected dose levels. These doses will be administered either as monotherapy or in combination with approved anti-cancer therapies, including pembrolizumab (200 mg IV every 3 weeks), or other standard-of-care therapies at the discretion of the site principal investigator (PI). Part B is enrolling approximately 140 subjects to further assess safety, tolerability, and preliminary efficacy at selected doses in expansion cohorts.

Subjects must have received standard of care (SOC) therapy for their advanced/metastatic tumors and subjects must have received, have been intolerant to, have been ineligible for, or have declined all treatment known to confer significant clinical benefit. Subjects must also have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST1.1), an Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2 and predicted life expectancy of greater than 3 months. An imaging scan is required at baseline, up to 28 days prior to treatment initiation. Subjects are required to provide an adequate tumor tissue sample (archival or fresh-tissue if no archival is available).

In all treatment arms, treatment continues until progressive disease (PD), unacceptable adverse events (AEs), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdrawal of consent, pregnancy of the subject, noncompliance with study dosing or procedure requirements, subject receiving approximately 2 years of RBS2418 monotherapy or combination therapy, or administrative reasons requiring cessation of treatment.

After the last dose of study drug, each subject will be followed for 30 days for AE monitoring. Serious adverse events (SAEs) will be collected for 90 days after the end of treatment or for 30 days after the end of treatment, if the subject initiates new anticancer therapy, whichever is earlier

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study. The subject may also provide consent for Future biomedical research (FBR). However, the subject may participate in the main study without participating in FBR.
2. 18 years of age on day of signing informed consent.
3. Male and female subjects with advanced unresectable, recurrent or metastatic tumors who have received standard of care (SOC) therapy for their advanced/metastatic tumors and have no other SOC therapy available. Additionally, subjects must have received, have been intolerant to, have been ineligible for, or have declined all SOC therapies known to confer significant clinical benefit.
4. Have histologically or cytologically confirmed cancer diagnosis based on pathology report.
5. Have a predicted life expectancy of greater or equal to 3 months.
6. Have measurable disease based on RECIST 1.1.
7. Have a performance status of 0, 1 or 2 using the ECOG Performance Scale within 14 days of first dose of study drug.
8. Willing to submit a pre-treatment (archival or fresh-tissue if no archival tissue is available) and on-treatment tissue sample. Subjects in whom the treating physician deems such biopsy is clinically contraindicated will be evaluated on a case-by-case basis for enrollment pending Sponsor consultation.

   Additionally, during the dose-escalation portion and if appropriate in the expansion phase of the study, the Sponsor may modify subject enrolment into various cohorts that have not begun enrolling yet such that ENPP1 and/or cGAS baseline expression level in the subject's tumor must be available and may guide enrolment eligibility for the study
9. Have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study drug (female subjects of childbearing potential who are not surgically sterilized or postmenopausal). If the urine test is positive, or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Demonstrate adequate organ function: hematological, renal, hepatic, coagulation parameters and obtained within 14 days prior to the first study treatment
11. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two highly effective contraceptive methods that result in a combined failure rate of < 1% per year during the treatment period and for at least 120 days after the last dose of study treatment or as instructed by the package insert of the chosen co-medication.
12. For male subjects: Agree that during the period specified above, men will not father a child. Male subjects must remain abstinent (refrain from heterosexual intercourse with women of childbearing potential), must be surgically sterile (e.g., vasectomy) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Use of any systemic anti-cancer therapy (including radiotherapy, chemotherapy, targeted therapy or immunotherapy) within 2 weeks prior to first dose of RBS2418 unless such therapy is being administered in combination with RBS2418 per protocol and has been approved by the Sponsor; or if subject has not recovered (i.e., Less than or equal to Grade 1 or returned to baseline level) from adverse events due to a previously administered agent; the following exceptions are allowed:

   * Palliative radiotherapy for bone metastases or soft tissue lesions should be completed > 7 days prior to baseline imaging
   * Hormone-replacement therapy or oral contraceptives
   * Subjects with Grade 2 neuropathy or Grade 2 alopecia
2. Subjects with evidence of rapid progression on prior therapy resulting in rapid clinical deterioration should be excluded from participation in the trial.
3. Currently participating and receiving trial therapy or has participated in a trial of an investigational agent and/or has used an investigational device within 28 days prior to Day 1.
4. Uncontrolled tumor-related pain
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
6. Malignancies other than indications open for enrollment within 3 years prior to Day 1, with the exception of those with negligible risk of metastasis or death treated with expected curative outcome, undergoing active surveillance or treatment-naïve for indolent tumors
7. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
8. Known hypersensitivity allergy or contraindication to any investigational product components administered as part of the combination therapy.
9. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
10. History or any evidence of interstitial lung disease
11. Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment.
12. Active HIV requiring therapy and Uncontrolled HIV*. HIV antibody testing recommended per investigator's clinical suspicion.
13. Active hepatitis B virus (HBV; hepatitis B surface antigen reactive) or active hepatitis C virus (HCV; qualitative RNA detected)*; such as requiring active therapy (e.g. subjects with a history of HCV are eligible as long as viral RNA is below level of detection); testing recommended per investigator's clinical suspicion.
14. Severe infections within 4 weeks prior to enrollment, including, but not limited to, hospitalization for complications of infection, bacteremia, or the presence of any active infection requiring systemic therapy.
15. Received therapeutic oral or IV antibiotics within 2 weeks prior to Day 1
16. History or current evidence of any condition, therapy, or laboratory abnormality that in the opinion of the treating investigator might confound the results of the trial or interfere with the subject's participation for the full duration of the trial.
17. Subjects with:

    * A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval of > 480 milliseconds (ms) (CTCAE Grade 1) using Fridericia's QT correction formula
    * A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
    * The use of concomitant medications that are known to prolong the QT/QTc interval unless there is evidence of the lack of QT/QTc interval prolongation at baseline.
18. Subjects with gastrointestinal disorders that may affect the absorption of the drug
19. Prior allogeneic stem cell or solid organ transplant.
20. Received a live, attenuated vaccine within 28 days prior to enrollment/cohort assignment or anticipation that such a live attenuated vaccine will be required during the trial
21. Known previous or ongoing, active psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Prisoner or subject who is compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infectious disease) illness.
23. Pregnant or lactating or intending to become pregnant or father children within the projected duration of the trial starting with the screening visit through 120 days after the last dose of pembrolizumab and/or RBS2418.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent dose limiting toxicities (DLT) | From 1- 21 days of the first cycle (each cycle is 21 days)
  When more than 1 DLT occurs in ≤ 6 patients in a dosing cohort, MTD has been exceeded and no more patients are to be treated at that dose level. No DLT observed at the highest dose level in Part A. Part A has been completed.
Peak plasma concentration (Cmax) of RBS2418 | Day 0 - 5
  maximum plasma concentration of RBS2418
Area under the plasma concentration versus time curve (AUC) | Day 0 - 5
  area under the curve for RBS2418
Optimal Biologically Active Dose (OBA) | Day 0 - 5
  Dose at which Ctrough plasma concentration of RBS2418 equal to or higher than ENPP1 EC90 in human serum is achieved. All dose levels (100-800 mg BID) achieved the endpoint. Part A has been completed.
Half-life (t1/2) | Day 0 - 5
  half-life of RBS2418
Number of participants with treatment emergent Adverse events | 30 days from last dose
  Adverse events, as graded by NCI CTCAE v5.0 including adverse events of special interest (AESI) classified by system organ class, preferred term, severity and relationship to drug

SECONDARY OUTCOMES:
Overall response rate (ORR) by RECIST | nine weeks from first dose
  Beginning with screening, all imaging assessments will be evaluated using RECIST 1.1. On- study imaging assessments will be performed Q9W. RECIST 1.1 will be used by the site for treatment decisions until the first radiographic evidence of PD.

CONTACTS AND LOCATIONS:
Overall Officials: Riboscience Chief Medical Officer, Study Director — Riboscience, LLC.
Locations (14):
- United States (14):
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Stanford Cancer Institute, Palo Alto, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Christiana Care Health Services, Newark, Delaware
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Tranquil Research, Webster, Texas
  - NEXT Virigina, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No